CLINICAL TRIAL: NCT02146521
Title: Prospective Study of Z-axis-limited Abdominal CT Guided by Region of Tenderness in the Diagnosis and Management of Adult Emergency Department Patients With Acute Nontraumatic Abdominal Pain and Tenderness
Brief Title: Limited Abdominal CT in ED Patients With Abdominal Pain
Acronym: LACTINEDAP
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050303
Record Dates: First submitted 2014-05-15; First posted 2014-05-26 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Abdominal Pain
Keywords: z-axis limited CT; computed tomography; CT; abdominal non-traumatic pain and tenderness; emergency patients
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients undergoing CT: Emergency department's patients undergoing CT scanning for evaluation of acute abdominal pain and tenderness

SUMMARY:
The purpose of the study is to compare the diagnosis and management (treatment and disposition) of adult emergency department patients with acute nontraumatic abdominal pain and tenderness, based on two CT techniques:

1. Standard (complete) abdominal-pelvic CT. The American College of Radiology calls for the cephalad limit of abdominal CT to begin at the dome of the diaphragm, and the caudad limit of pelvic CT to extend through the ischial tuberosities.
2. A z-axis restricted subset of images digitally obtained from the original CT dataset, determined by the region of tenderness identified by the examining emergency physician and marked on the patient prior to the performance of the CT. This z-axis restricted CT does not require any additional radiation exposure to the patient, as it will be produced by computer extraction of data from the original standard abdominal-pelvic CT.

The investigators hypothesize that the diagnosis and management will not differ when guided by the two CT scan interpretations. Radiation doses will be calculated for each of the two techniques.

DETAILED DESCRIPTION:
This will be a prospective study with informed consent from patient subjects.

Informed consent will be obtained prior to subject enrollment. The study protocol requires the following steps to be performed, each of which is described in more detail later in this document:

1. Potential patient subject is identified by research staff, by virtue of abdominal-pelvic CT being ordered for clinical evaluation of nontraumatic abdominal pain and tenderness, as determined by a board-certified attending emergency physician.
2. Research staff applies inclusion and exclusion criteria to confirm patient eligibility.
3. Potential subjects who fail one or more inclusion or meet one or more exclusion criteria are recorded in electronic research log with reason for exclusion but are not asked to participate in study. Recorded information includes age (if greater than 89, will simply be recorded as "greater than 89"), gender, race/ethnicity, date, and reason for exclusion. No identifiers are recorded for these patients. The purpose of this information is to allow comparison of the enrolled group with all patients with abdominal pain undergoing CT. This will be part of a CONSORT flow diagram, allowing readers to understand potential selection bias and to understand the probable clinical population in the context of all emergency department's (ED) patients undergoing abdominal CT.
4. Eligible potential subjects (meeting all inclusion and no exclusion criteria) are asked to participate in study with informed consent. The study will be introduced to potential subjects by the emergency physician caring for this patient. The study will be introduced only after CT for evaluation of abdominal pain and tenderness is ordered by the physicians caring for the patient, as this is a study inclusion criterion. Potential subjects who do not give informed consent to participate are recorded in electronic research log but not enrolled in study. No identifiers are recorded for these patients. Recorded information includes age (if greater than 89, will simply be recorded as "greater than 89"), gender, race/ethnicity, date, and reason for exclusion. No identifiers are recorded for these patients.
5. Patients who give informed consent are enrolled in study as subjects.
6. Attending board-certified emergency physician places skin surface markers delineating region of abdominal tenderness, using an examination technique described below. Patient is marked with stickers while in supine position with arms above head, as required for CT. Attending board-certified emergency physician also places additional markers to blind radiological interpretation with respect to actual area of tenderness. Attending board-certified emergency physician is also asked to report the working diagnosis, treatment and disposition plan prior to CT scan being performed. An electronic standardized reporting form will be used. Reporting forms are designed in a format of electronic surveys and will be stored on password-protected server, designed specifically for research purposes. The information to be collected will be the same as the information in the attached appendices.
7. Patient undergoes CT scan of complete abdomen and pelvis following usual institutional protocol, concordant with American College of Radiology standard.1
8. Images corresponding to the region of tenderness (z-axis restricted) are loaded onto a server. A board-certified attending radiologist blinded to the remaining CT images interprets the z-axis limited CT images and generates an electronic report, using a standardized research reporting system. The report is electronically time-stamped and cannot be altered.
9. The attending board-certified emergency physician is immediately provided with the electronic CT report from the z-axis limited CT. That physician immediately completes a standardized electronic research reporting form, indicating the current clinical diagnosis, treatment plan, and disposition. The form is electronically time-stamped and cannot be altered.
10. The board-certified attending radiologist who interpreted the z-axis restricted CT is then immediately contacted and interprets the complete CT, including all available images. A report is generated using similar standardized electronic research reporting system used for the z-axis restricted CT. The report is electronically time-stamped and cannot be altered.
11. The attending board-certified emergency physician is immediately provided with the CT report from the complete CT. That physician immediately completes an electronic standardized research reporting form, indicating the current clinical diagnosis, treatment plan, and disposition. The form is electronically time-stamped and cannot be altered.
12. Patient care then proceeds according to the usual clinical standard in the institution.
13. Subject records are reviewed to determine final diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* emergency department's patients undergoing CT evaluation for acute abdominal pain and tenderness (acute is defined as onset of current episode within 7 days of emergency department presentation).

Exclusion Criteria:

* neurological disorders
* altered mental status
* history of intra-abdominal surgery in the past 30 days
* BMI higher than 35
* immunocompromised patients
* abdominal trauma in the past 30 days
* CT is ordered for the following indications:
* isolated vomiting
* fever without source
* staging of malignancy
* isolated flank pain or suspected renal colic

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of the emergency department undergoing CT evaluation for acute abdominal pain and tenderness
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis, treatment and disposition | Records will be reviewed from the ED visit date to the date of discharge from the hospital or up to 30 days following ED visit, whichever comes last
  The diagnosis, treatment, and disposition plans based on the z-axis restricted CT and the full CT will be compared for agreement.

SECONDARY OUTCOMES:
radiation reduction | Records will be reviewed 30 days after the ED visit or date of discharge from the hospital, whichever comes first
  The radiation doses resulting from a z-axis restricted CT and the full CT will be compared using dose-length products.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua S Broder, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States